CLINICAL TRIAL: NCT05857618
Title: A Survey and Chart Review to Determine if Patients Exposed to General Anesthesia Significant Numbers of Times Would Increase the Risk for Intraoperative Awareness With Explicit Recall.
Brief Title: Study to Determine if Patients Exposed to General Anesthesia Significant Numbers of Times Would Increase the Risk for Intraoperative Awareness.
Acronym: EXPLICIT-RCL
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 17-0929
Record Dates: First submitted 2022-11-18; First posted 2023-05-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-07

CONDITIONS: Intraoperative Awareness; General Anesthesia
Keywords: explicit recall; Intraoperative; Intraoperative awareness; General Anesthesia; Intraoperative recall
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have undergone exposer to General Anesthesia: Patients who have undergone general anesthesia at the University of Chicago Medical Center more than 20 times or patients who have general anesthesia 5 or fewer times in the past.

SUMMARY:
This study will detect whether prior exposure to general anesthesia multiple times is associated with an increased incidence of awareness with explicit recall (AWR). This is especially important because patients who need to undergo multiple events of general anesthesia are medically some of the most vulnerable populations. The study hypothesizes that patients with significant exposure to general anesthesia have a higher incidence of AWR. This study may help clinicians and patients to better understand how to manage anesthesia care so that the safety and comfort of patients can be improved.

DETAILED DESCRIPTION:
Each year, tens of millions of Americans undergo general anesthesia. One of the biggest fears patients have regarding general anesthesia is experiencing intraoperative awareness. That means that the patients "wake" during surgery and become aware of their environment. Prior studies have shown that intraoperative awareness with explicit recall (AWR) occurs in 0.1%-0.2% of patients undergoing general anesthesia. Patients have reported different forms of AWR, including feeling the sensation of pain, difficulty breathing, or recalling conversations. AWR can leave a lasting negative effect on patients. In one study, 56.3% of patients who experienced AWR met the diagnostic criteria for PTSD with functional impairment. Another study found that PTSD was experienced by as many as 70% of patients who had AWR.5 These patients fear undergoing further medical treatment requiring anesthesia and suffer quality of life issues related to their episode(s) of AWR. The goal of this study is to determine whether there is a particular group of patients, those that have been anesthetized many times, at high risk for AWR and then to design protocols to prevent this from happening.

Rationale for Conducting this Research

While the incidence of intraoperative awareness with explicit recall (AWR) is 0.1%-0.2% in general population undergoing general anesthesia, higher incidence has been reported in the populations with special risk factors, such as obstetric, cardiac and trauma surgeries. Patients with a history of awareness are at increased risk of intraoperative awareness. However, it is not certain whether this association is related to the number of anesthesia exposure or the development of resistance to anesthetics in these patients. Prior studies have demonstrated that the incidence of AWR in females is threefold higher than in males and that AWR is higher in patients with difficult airways and in patients with drug addiction. In addition, patients with an ASA Status of III-V had a greater than 2.4 odd of AWR than patients with an ASA Status of I-II. Most recently, we took care of two young adult patients who had more than 20 surgeries requiring general anesthesia since their childhood and reported multiple incidents of AWR. One of patients had a new episode of AWR during a regular surgery a few months ago despite extra measures were taken by her anesthesiologists. In addition, we found animals that were anesthetized multiple times showed change in their sensitivity to general anesthetics. To date, there has not been a study that has looked at whether patients who have undergone general anesthesia a significant number of times (n>20) have a higher incidence of AWR.

Primary Objective

To determine whether patients who have undergone general anesthesia significant number of times have a significantly higher incidence of intraoperative awareness with explicit recall (AWR) as compared to the general population.

Secondary Objective Allows us to better understand the cause of AWR in this population. It may help us to improve clinical care and comfort for patients who are at a higher risk for intraoperative awareness.

Patients that meet the eligibility criteria will be contacted by phone to provide consent to participate in the study. Patients who refuse to consent will not be included in the study and that data will not be saved. Of the patients who consent, a standardized phone interview by trained interviewers will be carried out and this data will be collected and stored in an encrypted computer hard drive. This data will be reviewed by anesthesiologists using a standard criteria to elucidate whether the patient experienced intraoperative awareness with explicit recall. The questionnaire includes the common complaints from the report of a North American anesthesia awareness registry. In addition to the questionnaire, the study team will perform a chart review on eligible patients collecting data on thier medical and surgical history, current medications and clinical situations when AWR occurred.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been exposed to general anesthesia greater than 20 times or who have been exposed to general anesthesia 5 or fewer times between January 1, 1985 and June 15, 2017
* Patients/their Guardians who consent to participate in the study.
* Patients for whom a determination of AWR status can be made by anesthesiologists based on a standardized criteria.
* Must be at least 7 years of age or older.

Exclusion Criteria:

* Healthy volunteers,
* Patients who cannot recall whether or not they have experienced intraoperative awareness with explicit recall

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the University of Chicago Medical Center who are 7 years or older who have been exposed to general anesthesia either less than 5 times or greater than 20 times.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Awareness with Explicit Recall for patients who underwent more than 20 general anesthesia events | Until study completion; up to 1 year.
  The Number of incidences of intraoperative awareness with explicit recall with patients undergoing general anesthesia greater than 20 times using the 5-question modified Brice questionnaire

SECONDARY OUTCOMES:
Intraoperative Awareness with Explicit Recall for patients who underwent less than 5 general surgeries involving general anesthesia | Until study completion; up to 1 year.
  The Number of incidences of intraoperative awareness with explicit recall with patients undergoing general anesthesia less than 5 times using the 5-question modified Brice questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No